CLINICAL TRIAL: NCT05881798
Title: Post-Market Celect Platinum Vena Cava Filter and Günther Tulip Retrieval Set Study
Brief Title: Post-Market Celect Platinum Vena Cava Filter and Gunther Tulip Retrieval Set Study
Status: Recruiting | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: MDR-2126
Record Dates: First submitted 2023-05-02; First posted 2023-05-31 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Deep Vein Thrombosis; Venous Thromboembolism; Pulmonary Embolism
Keywords: Celect Platinum Vena Cava Filter; Gunther Tulip Vena Cava Filter Retrieval Set
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients indicated for the placement of a Celect Platinum Vena Cava Filter: Patients indicated for the placement of a Celect Platinum Vena Cava Filter
  Interventions: Device: Celect Platinum Vena Cava Filter

INTERVENTIONS:
Device: Celect Platinum Vena Cava Filter — Inferior vena cava filter

SUMMARY:
This prospective, observational, post-market study will be performed to collect patient-level data on the Celect Platinum Vena Cava Filter Sets and the Günther Tulip Vena Cava Filter Retrieval Set to confirm continued safety and performance of the devices throughout their expected lifetime and continued acceptability of the benefit:risk ratio. Additionally, the study intends to evaluate longer-term (i.e., up to 5 years) outcome data while the filter is indwelling.

ELIGIBILITY:
Inclusion Criteria:

* A patient dataset is deemed suitable for inclusion if the patient has a procedure where a Celect Platinum Vena Cava Filter is placed
* Subject has not previously participated in the Cook MDR-2126 study.

Exclusion Criteria:

* Patients will be excluded from enrollment if the patient or his/her legally authorized representative objects to collection and processing of his/her data or is not willing to sign the Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient dataset is deemed suitable for inclusion in the study if the patient has a procedure where a Celect Platinum Vena Cava Filter
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Filter-related primary endpoint (safety) | Index procedure through 12-months post procedure
  Freedom from major adverse events through 12 months (365 ± 30 days), defined as clinically significant IVC penetration, migration of filter (>2 cm)/filter components, filter fracture, embolization of filter or filter fragments to the heart or lungs, IVC thrombotic occlusion, symptomatic deep vein thrombosis while a filter is indwelling, access site complications with clinical sequelae, and procedure/device-related death.
Filter-related primary endpoint (performance) | 12-months post procedure
  Performance:
  Technical placement success and freedom from symptomatic PE while a filter is indwelling through 12 months (365 ± 30 days).These values will be reported as aggregate. Technical placement success - Deployment of filter in a location suitable to provide sufficient mechanical protection against PE with no filter deformation, fracture, premature release, or clinical migration.
Filter Retrieval-related primary endpoint | Through 30-days post procedure
  Freedom from major adverse events through 30 days post-procedure, defined as access site complications with clinical sequelae, and procedure/device-related death.
Filter Retrieval-related primary endpoint | At the time of retrieval procedure
  Technical retrieval success, defined as endovascular retrieval of complete filter.

CONTACTS AND LOCATIONS:
Locations (2):
- Parc Tauli, Sabadell, Spain
- Royal Liverpool Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request immediately after approval or clearance of the product and ending 5 years after approval or clearance. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.